CLINICAL TRIAL: NCT02206854
Title: Bioavailability, Pharmacokinetics and Tissue Distribution of R-flurbiprofen Capsules in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gerd Geisslinger (Other)
Collaborators: Fraunhofer Institute for Translational Medicine and Pharmacology ITMP (Other)
Responsible Party: Sponsor-Investigator, Gerd Geisslinger, Professor Dr. Dr. Gerd Geisslinger, Goethe University
Organization: Goethe University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: FLIP0112; 2012-001425-27 (EudraCT Number)
Record Dates: First submitted 2014-07-31; First posted 2014-08-01 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Volunteers
Keywords: Pharmakokinetic; capsules; R-Flurbiprofen
MeSH Terms: interventions — tarenflurbil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- R-flurbiprofen (Experimental): 200 mg R-flurbiprofen in gelatine capsules once
  Interventions: Drug: R-flurbiprofen

INTERVENTIONS:
Drug: R-flurbiprofen — 200 mg gelatine capsule once orally
  Other Names: Tarenflurbil

SUMMARY:
For previous clinical trials, R-flurbiprofen has been prepared in tablet form. In this study R-flurbiprofen, will be available as gelatine capsules.

This study aims to show the bioavailability of R-flurbiprofen when administered in gelatine capsules. The serum availability will be determined by analysis of pharmakokinetic (pK)-blood samples at different time points. To assess the safety of the administered capsules adverse events will be documented.

Analysis of lipid signaling molecules in plasma will be done to assess the role of this molecules as variable for therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18 to 65 years
* Body mass index (BMI) between 18.5 und 30 kg/m2
* Subject is judged to be in good health based on medical history, physical examination, vital sign measurements, and laboratory safety tests
* Subject has no evidence of clinically significant abnormality on echocardiogram (ECG) performed at screening visit and/or prior to administration of the study drug
* Non-Smoker
* Subjects providing informed consent

Exclusion Criteria:

* Subjects with known hypersensitivity to study medication
* Subjects who have experienced asthma, urticaria, or allergic-type reactions after taking aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs)
* Subjects with a history of peptic ulcer disease and/or gastrointestinal bleeding
* Pregnant women (pregnancy rapid assay required for women with childbearing potential), women currently breast-feeding, or with the intention to breast-feed
* History or evidence of active malignancy within the 24 months prior to entry.
* Subject has a history of fainting during blood draws.
* Subject has had major surgery, donated or lost 1 unit of blood (approximately 500 ml) in the last 4 weeks
* Subject is currently a regular user (including "recreational use) of illicit drugs or has a history of drug (including alcohol) abuse within approximately 2 years.
* Active or history of drug abuse,
* Chronic or acute renal, hepatic or metabolic disorder
* Participation in a clinical study within 30 days prior to screening
* Subjects with immunodeficiencies such as established acquired immunodeficiency syndrome.
* Subject is unable to refrain from or anticipates the use of any medication, (including prescription and non-prescription drugs or herbal remedies (such as St. John's Wort) beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study drug until the follow-up visit.
* Subject has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
* There is any concern of the investigator regarding the safe participation of the subject in the study or for any other reason, the investigator considers the subject inappropriate for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) | prior to administration, 30, 60, 90, 120 and 150 minutes and 3, 4, 5, 6, 8, 10, 12 and 24 hours after administration
  assessment of concentration at baseline (0), 30, 60, 90, 120 and 150 minutes and 3, 4, 5, 6, 8, 10, 12 and 24 hours after administration of study medication
Time to maximum concentration (Tmax; hours) | prior to administration, 30, 60, 90, 120 and 150 minutes and 3, 4, 5, 6, 8, 10, 12 and 24 hours after administration
Maximum concentration (Cmax). | prior to administration, 30, 60, 90, 120 and 150 minutes and 3, 4, 5, 6, 8, 10, 12 and 24 hours after administration
Terminal elimination half-life (t1/2) | prior to administration, 30, 60, 90, 120 and 150 minutes and 3, 4, 5, 6, 8, 10, 12 and 24 hours after administration

SECONDARY OUTCOMES:
Number of volunteers with serious and Non serious adverse events | Up to day 15
  Number and type of Adverse Events (AEs) and Serious Adverse Events (SAEs) will be documented at V1 (predose and after administration) and at V3 (follow-up visit 8 to 15 days after administration of study medication)
Analysis of plasma lipid profile | prior and 30, 60, 90, 120 and 150 minutes and 3, 4, 5, 6, 8, 10, 12 and 24 hours after administration
  parallel to pK-Analysis plasma lipid profile will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Geisslinger, Prof MD, Principal Investigator — Goethe University
Locations (1):
- Johann Wolfgang Goethe University Hospital, Frankfurt, Germany